CLINICAL TRIAL: NCT07034690
Title: A Prospective, Type I Hybrid Effectiveness-implementation, Open Label, Randomized Study to Evaluate the Impact of a Targeted Lipid Optimization Program on LDL-C Control in at- Risk Adult Patients From Abu Dhabi, United Arab Emirates (UAE) With Dyslipidemia
Brief Title: Study to Evaluate the Impact of a Targeted Lipid Optimization Program on LDL-C Control in At-risk Adult Patients With Dyslipidemia
Acronym: OPTIMA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CKJX839A1AE02
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Dyslipidemia,; ASCVD,; lipid optimization program,; LDL-C target,; educational intervention,; hybrid effectiveness-implementation study
MeSH Terms: conditions — Atherosclerosis; Dyslipidemias | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Participants receive Health Education Intervention alongside standard of care
  Interventions: Other: Educational Material; Other: Standard of care
- Control Group (Other): Participants receive Standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Educational Material — Health Education Intervention delivered via clinic visits (every 4 months) and virtual sessions (between each clinic visit)
  Arms: Intervention group
Other: Standard of care — Standard of care

SUMMARY:
This study is an open label, randomized, prospective, type I hybrid effectiveness- implementation, pragmatic clinical trial to evaluate the impact of a targeted lipid optimization program on LDL-C control in participants with dyslipidemia who are at high risk or very high risk of cardiovascular events.

DETAILED DESCRIPTION:
The treatment of interest is a lipid optimization program in the form of a health education intervention delivered via clinic visits (every 4 months) and virtual sessions (between each clinic visit).

No active drug treatment will be provided. The intervention in this study will involve the implementation of a lipid optimization, education program for patients at high risk and very high risk of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ASCVD (coronary heart disease, peripheral arterial disease and/or cerebrovascular disease)
* High risk or very high risk for cardiovascular events (as per the 2019 ESC/EAS guidelines [1] for the management of dyslipidemias)
* Lipid levels:

  * High risk: LDL-C ≥70 mg/dl (or > 1.8 mmol/L) or non-HDL-C ≥100 mg/dl
  * Very high risk: LDL-C ≥55 mg/dl (or > 1.4 mmol/L) or non-HDL-C ≥85 mg/dl
* Male or Female
* 18 years or older
* Seen by a specialist who is prescribing advanced lipid lowering treatments (LLTs) (cardiologist, endocrinologist or any other relevant specialist)
* Currently taking maximum-tolerated statins
* Ability to participate in educational program (must be able to watch online videos)
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Any surgical or medical condition, which in the opinion of the Investigator, may place the participant at higher risk from his/her participation in the study, or is likely to prevent the participant from complying with the requirements of the study or completing the study.
* Unwillingness or inability (e.g., physical or cognitive) to comply with study procedures (including adherence to study visits).
* Participation in any other interventional study.
* Inability to travel to study sites for in-person clinic visits.
* Responsible physician clinical decision not to engage the identified patient.
* Refusal of the potential participant to sign the consent and be included in the model.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving target LDL-C goals based on CV risk | Baseline, month 12
  Percentage of participants achieving target Low-Density Lipoprotein Cholesterol (LDL-C) goals based on Cardiovascular (CV) risk stratified by group:
  * Very high risk: <55 mg/dl
  * High risk: <70 mg/dl

SECONDARY OUTCOMES:
Percentage of participants achieving or maintaining target LDL-C goals based on CV risk | Baseline, month 24
  Percentage of participants achieving or maintaining target Low-Density Lipoprotein Cholesterol (LDL-C) goals based on Cardiovascular (CV) risk stratified by group:
  * Very high risk: <55 mg/dl
  * High risk: <70 mg/dl
Change of LDL-C | Baseline, month 12 and month 24
  Change of Low-Density Lipoprotein Cholesterol (LDL-C) from baseline at 12 months and 24 months in both study groups
Change in the proportion of participants receiving advanced lipid lowering therapies | Month 12 and Month 24
  Change in the proportion of participants receiving advanced lipid lowering therapies at 12 months and 24 months from baseline, for each group
Proportion of participants from the intervention group who complete all visits | 24 months
  Proportion of participants from the intervention group who complete all:
  * In clinic visits
  * Virtual sessions
Proportion of participants from the intervention group who discontinue the education program | 12 months
  Proportion of participants from the intervention group who discontinue the education program before the 12 month study visit
Proportion of days covered | Baseline, month 12 and month 24
  Proportion of days covered (for statins and non-statin lipid therapies)
Number of hospitalizations | 24 months
  Number of hospitalizations during the 12 month active intervention period and the 12 month follow up period
Number of outpatient visits | 24 months
  Number of outpatient visits during the 12 month active intervention period and the 12 month follow up period
Number of ER visits | 24 months
  Number of Emergency Room (ER) visits during the 12 month active intervention period and the 12 month follow up period
Associated costs | 24 months
  Associated costs during the 12 month active intervention period and the 12 month follow up period
Number of LDL-C tests performed | 24 months
  Number of Low-Density Lipoprotein Cholesterol (LDL-C) tests performed, analyzed according to:
  * Site (clinic)
  * Healthcare Professional (HCP) specialty (Cardiologists, Endocrinologists, internist, etc.)
  * Baseline characteristics (e.g. age, sex, ethnicity, Cardiovascular risk status)
Change in knowledge awareness scores: | Baseline, month 12 and month 24
  Awareness regarding lipid management amongst those participants in the intervention group will be measured using a knowledge awareness questionnaire. The same questionnaire will be administered at baseline, 12 months and 24 months, enabling scores to be compared across the study duration.
  The knowledge awareness questionnaire scale has a minimum score of 0 and maximum score of 17 points. A high score will indicate higher participant awareness.
Change in WHO BREF quality of life scores | Baseline, month 12 and month 24
  WHO BREF questionnaire assesses QoL across four main domains: physical health, psychological health, social relationships, and environmental health.
  Participants will respond to each item using a Likert scale (ranging from 1 to 5) indicating their level of agreement or satisfaction. Higher scores typically indicate better QoL.
Qualitative surveys among focus groups of HCPs and participants to evaluate implementation outcomes | month 12 and month 24
  Implementability of the lipid optimization program will be assessed during focus group sessions that explore satisfaction, costs, and acceptance of the program from the perspective of HCPs and participants

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com